CLINICAL TRIAL: NCT04194944
Title: LIBRETTO-431: A Multicenter, Randomized, Open-Label, Phase 3 Trial Comparing Selpercatinib to Platinum-Based and Pemetrexed Therapy With or Without Pembrolizumab as Initial Treatment of Advanced or Metastatic RET Fusion-Positive Non-Small Cell Lung Cancer
Brief Title: A Study of Selpercatinib (LY3527723) in Participants With Advanced or Metastatic RET Fusion-Positive Non-Small Cell Lung Cancer
Acronym: LIBRETTO-431
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17479; J2G-MC-JZJC (Other: Eli Lilly and Company); 2019-001979-36 (EudraCT Number)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: targeted therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — selpercatinib; Carboplatin; Cisplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Selpercatinib - Treatment A (TRT A) (Experimental): 160 milligram (mg) Selpercatinib administered orally twice daily (BID) continuously in 21-day cycles.
  Interventions: Drug: Selpercatinib
- Pemetrexed and Platinum with or without Pembrolizumab - (TRT B) (Active Comparator): Pemetrexed 500 milligrams per meter squared (mg/m2) administered intravenously (IV) on Day 1, every 3 weeks (Q3W), plus investigator's choice of carboplatin area under the concentration versus time curve 5 (AUC 5 [maximum dose of 750 mg] IV), or cisplatin (75 mg/m2 cisplatin IV) on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292
  Arms: Selpercatinib - Treatment A (TRT A)
Drug: Carboplatin — Administered IV
  Arms: Pemetrexed and Platinum with or without Pembrolizumab - (TRT B)
Drug: Cisplatin — Administered IV
  Arms: Pemetrexed and Platinum with or without Pembrolizumab - (TRT B)
Drug: Pemetrexed — Administered IV
  Arms: Pemetrexed and Platinum with or without Pembrolizumab - (TRT B)
Drug: Pembrolizumab — Administered IV
  Arms: Pemetrexed and Platinum with or without Pembrolizumab - (TRT B)

SUMMARY:
The reason for this study is to see if the study drug selpercatinib compared to a standard treatment is effective and safe in participants with rearranged during transfection (RET) fusion-positive non-squamous non-small cell lung cancer (NSCLC) that has spread to other parts of the body. Participants who are assigned to the standard treatment and discontinue due to progressive disease have the option to potentially crossover to selpercatinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, Stage IIIB-IIIC or Stage IV non-squamous NSCLC that is not suitable for radical surgery or radiation therapy.
* A RET gene fusion in tumor and/or blood from a qualified laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate hematologic, hepatic and renal function.
* Willingness of men and women of reproductive potential to observe conventional and highly effective birth control for the duration of treatment and for 6 months after.
* Ability to swallow capsules.

Exclusion Criteria:

* Additional validated oncogenic drivers in NSCLC if known.
* Prior systemic therapy for metastatic disease. Treatment (chemotherapy, immunotherapy, or biological therapy) in the adjuvant/neoadjuvant setting is permitted if it was completed at least 6 months prior to randomization.
* Major surgery within 3 weeks prior to planned start of selpercatinib.
* Radiotherapy for palliation within 1 week of the first dose of study treatment or any radiotherapy within 6 months prior to the first dose of study treatment if more than 30 Gy to the lung.
* Symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or untreated spinal cord compression.
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of selpercatinib or prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 milliseconds.
* Active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing intercurrent illness, such as hypertension or diabetes, despite optimal treatment.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.
* Pregnancy or lactation.
* Other malignancy unless nonmelanoma skin cancer, carcinoma in situ of the cervix or other in situ cancers or a malignancy diagnosed ≥2 years previously and not currently active.
* Uncontrolled, disease related pericardial effusion or pleural effusion.
* Requiring chronic treatment with steroids.

Exclusion Criteria for Participants Receiving Pembrolizumab:

* History of interstitial lung disease or interstitial pneumonitis.
* Active autoimmune disease or any illness or treatment that could compromise the immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2030-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (196):
- Argentina (5):
  - Centro de Oncología e Investigación de Buenos Aires, Berazategui, Buenos Aires
  - Fundacion CENIT para la Investigacion en Neurociencias, Caba, Buenos Aires
  - Clinica Viedma, Viedma, Río Negro Province
  - Alexander Fleming, Ciudad de Buenos Aires
  - Clínica El Castaño, San Juan
- Australia (7):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Peninsula Oncology Centre, Frankston
- Belgium (7):
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Delta, Roeselare, West Flanders
  - UZ Gent Hospital, Ghent
  - AZ Sint-Maarten, Campus Leopoldstraat 2, Mechelen
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (11):
  - Hospital Sírio Libanês, São Paulo, Brazil
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital de Cancer de Londrina, Londrina, Paraná
  - Grupo COI - Clínicas Oncológicas Integradas, Rio de Janeiro, Rio de Janeiro
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Sírio Libanês, São Paulo
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (15):
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - First affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou
  - Shanghai Chest Hospital, Shanghai
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava - Vitkovice
  - Fakultni nemocnice Bulovka, Prague
- France (6):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Institut Régional du Cancer Montpellier, Montpellier, Hérault
  - Chu Grenoble Alpes, La Tronche, Isère
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand, Puy-de-Dôme
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
- Germany (8):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Klinikverbund Kempten-Oberallgäu, Immenstadt im Allgäu, Bavaria
  - Franziskus-Hospital Harderberg, Georgsmarienhütte, Lower Saxony
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
- Greece (4):
  - Sotiria Thoracic Diseases Hospital of Athens, Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Krítí
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - G. Papanikolaou General Hospital, Thessaloniki, Thessaloníki
- Hong Kong (2):
  - Hong Kong United Oncology Centre, Jordan, Kowloon
  - Prince of Wales Hospital, Shatin
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Rambam Health Care Campus, Haifa, Ḥeifā
- Italy (13):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - Ospedale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Ospedale San Gerardo-ASST Monza, Monza, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Humanitas, Rozzano, Milano
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Torino
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - IRCCS - AOU di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena, Roma
- Japan (11):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Kindai University Hospital- Osakasayama Campus, Osaka Sayama-shi, Osaka
  - Tominaga Hospital, Nakatogari, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
- Mexico (3):
  - Health Pharma Professional Research S.A. de C.V:, Mexico City, Federal District
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara, Jalisco
  - Oncologico Potosino, S.C., San Luis Potosí City
- Netherlands (4):
  - Ziekenhuis St. Jansdal, Harderwijk, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Amsterdam UMC, locatie VUmc, Amsterdam
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Romania (7):
  - Gral Medical Diagnostic Center, Bucharest, București
  - Institutul Oncologic, Bucharest, București
  - Constanta County Emergency Clinical Hospital Sf.Ap.Andrei, Constanța, Constanța County
  - Cabinet Medical Oncomed, Timișoara, Timiș County
  - Spitalul Universitar de Urgență București, Bucharest
  - Institutul Oncologic, Cluj-Napoca
  - Spitalul Județean Sfântul Ioan cel Nou Suceava, Suceava
- Russia (10):
  - GBUZ Republican Clinical Oncological Dispensary, Ufa, Baškortostan, Respublika
  - Kaluga Regional Clinical Oncology Center, Kaluga, Kalužskaja Oblast
  - Murmansk Regional Clinical Hospital P.A. Bayandina, Murmansk, Murmansk Oblast
  - Samara Regional Clinical Oncology Center, Samara, Samara Oblast
  - Saint-Petersburg Scientific-Practical Center of Specialized Kinds of Medical Care (oncological) named afte -T, Saint Petersburg, Sankt-Peterburg
  - Scientific research institution of oncology named after N.N. Petrov, Saint Petersburg, Sankt-Peterburg
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Republican Clinical Oncology Dispensary, Kazan'
  - First Moscow State Medical University I.M. Sechenov, Moscow
  - Hadassah Medical, Moscow
- Tan Tock Seng Hospital, Singapore, Singapore
- South Korea (9):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Korea
  - Asan Medical Center, Seoul, Korea
  - Gyeongsang National University Hospital, Jinju, Kyǒngsangnam-do
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Boramae Medical Center, Dongjak-gu, Seoul-teukbyeolsi [Seoul]
  - Konyang University Hospital, Daejeon
  - Samsung Medical Center, Seoul
- Spain (23):
  - Hospital Fundacion Son Llatzer, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [Barcelona]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, Galicia [Galicia]
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (14):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Buddhist Dalin Tzu Chi General Hospital, Dalin Town, Chiayi
  - Chang Gung Memorial Hospital - Linkou, Guei Shan Township, Taoyuan County
  - E-Da hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - Tri-Service General Hospital, Neihu Taipei
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (12):
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Abdurrahman Yurtaslan Ankara Oncology, education and Research Hospital, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Memorial Antalya Hastanesi, Antalya
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - Istanbul Medeniyet University, Istanbul
  - zmir Katip Çelebi Üniversitesi Atatürk Eitim Ve Aratrma Hastanesi, Izmir
  - Izmir Medical Park Hospital, Izmir
  - Inonu Universitesi Turgut Ozal Tıp Merkezi, Malatya
  - Acıbadem Maslak Hastanesi, Sarıyer
- Ukraine (11):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, "Dnipro State Medical University", Dnipro, Dnipropetrovsk Oblast
  - CNPE "Regional Center of Oncology", Kharkiv, Kharkivs’ka Oblast’
  - Odessa Regional Oncology Center, Odesa, Odesa Oblast
  - Sumy regional clinical oncological dispensary, Sumy, Sumska Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council", Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "Volyn Regional Medical Oncology Centre" of the Volyn Regional Council, Lutsk, Volyn Oblast
  - "Oncolife" LLC, Zaporizhya, Zaporizhzhia Oblast
  - Regional Municipal Non-profit Enterprise "Bukovinian Clinical Oncology Center", Chernivtsi
  - Medical Center "Mriya Med-Service", LLC, Kryvyi Rig
  - Municipal non-profit enterprise "Kyiv City Clinical Oncology Center" of executive body of Kyiv City Counci -T, Kyiv
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa
- City Hospital, Nottingham University Hospitals, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Perol M, Solomon BJ, Goto K, Park K, Nadal E, Bria E, Martin C, Bar J, Williams JN, Puri T, Li J, Uh MK, Lin BK, Zhou C. CNS Protective Effect of Selpercatinib in First-Line RET Fusion-Positive Advanced Non-Small Cell Lung Cancer. J Clin Oncol. 2024 Jul 20;42(21):2500-2505. doi: 10.1200/JCO.24.00724. Epub 2024 Jun 3. PMID 38828957
- [Derived] Zhou C, Solomon B, Loong HH, Park K, Perol M, Arriola E, Novello S, Han B, Zhou J, Ardizzoni A, Mak MP, Santini FC, Elamin YY, Drilon A, Wolf J, Payakachat N, Uh MK, Rajakumar D, Han H, Puri T, Soldatenkova V, Lin AB, Lin BK, Goto K; LIBRETTO-431 Trial Investigators. First-Line Selpercatinib or Chemotherapy and Pembrolizumab in RET Fusion-Positive NSCLC. N Engl J Med. 2023 Nov 16;389(20):1839-1850. doi: 10.1056/NEJMoa2309457. Epub 2023 Oct 21. PMID 37870973
- [Derived] Claerhout S, Lehnert S, Vander Borght S, Spans L, Dooms C, Wauters E, Vansteenkiste J, Weynand B, Deraedt K, Bourgain C, Vanden Bempt I. Targeted RNA sequencing for upfront analysis of actionable driver alterations in non-small cell lung cancer. Lung Cancer. 2022 Apr;166:242-249. doi: 10.1016/j.lungcan.2022.02.013. Epub 2022 Mar 1. PMID 35378489
- [Derived] Solomon BJ, Zhou CC, Drilon A, Park K, Wolf J, Elamin Y, Davis HM, Soldatenkova V, Sashegyi A, Lin AB, Lin BK, F Loong HH, Novello S, Arriola E, Perol M, Goto K, Santini FC. Phase III study of selpercatinib versus chemotherapy +/- pembrolizumab in untreated RET positive non-small-cell lung cancer. Future Oncol. 2021 Mar;17(7):763-773. doi: 10.2217/fon-2020-0935. Epub 2020 Nov 5. PMID 33150799
- See also: A Study of Selpercatinib (LY3527723) in Participants With Advanced or Metastatic RET Fusion-Positive Non-Small Cell Lung Cancer — https://trials.lilly.com/en-US/trial/230195

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If a participant has a recorded death on study, or is alive and being followed but off treatment, then the participant can be considered to be study completer.
Groups:
- Selpercatinib (TRT A): 160 milligram (mg) Selpercatinib administered orally, twice daily (BID) continuously in 21-day cycles.
- Pemetrexed and Platinum With or Without Pembrolizumab (TRT B): Pemetrexed 500 milligrams per meter squared (mg/m2) administered intravenously (IV) on Day 1, every 3 weeks (Q3W), plus investigator's choice of carboplatin area under the concentration versus time curve 5 (AUC 5 [maximum dose 750 mg]) IV, or cisplatin 75mg/m2 IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Period: Overall Study
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Started | 159 | 102
Received at Least One Dose of Study Drug | 158 | 98
Completed | 61 | 70
Not Completed | 98 | 32
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — On Treatment | 93 | 30

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT): All randomized participants, even if a participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Groups:
- Selpercatinib (TRT A): 160 mg Selpercatinib administered orally BID continuously in 21-day cycles.
- Pemetrexed and Platinum With or Without Pembrolizumab (TRT B): Pemetrexed 500 mg/m2, IV on Day 1 Q3W plus investigator's choice of carboplatin (AUC 5 [maximum dose 750 mg] IV) or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
- Total: Total of all reporting groups
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B) | Total
Number analyzed (Participants) | 159 | 102 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.3) | 60.8 (11.4) | 60.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 57 | 143
  Male | 73 | 45 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 92 | 52 | 144
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 58 | 43 | 101
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 4 | 1 | 5
  Czechia | 0 | 1 | 1
  Russia | 1 | 2 | 3
  Greece | 2 | 0 | 2
  Netherlands | 2 | 1 | 3
  South Korea | 8 | 8 | 16
  China | 62 | 28 | 90
  Brazil | 7 | 1 | 8
  Poland | 0 | 1 | 1
  France | 2 | 4 | 6
  Argentina | 2 | 0 | 2
  Japan | 15 | 10 | 25
  Ukraine | 0 | 5 | 5
  Spain | 7 | 9 | 16
  Canada | 2 | 1 | 3
  Turkey | 8 | 0 | 8
  Belgium | 3 | 3 | 6
  Taiwan | 2 | 4 | 6
  Italy | 20 | 12 | 32
  Mexico | 4 | 1 | 5
  Israel | 1 | 4 | 5
  Australia | 2 | 2 | 4
  Germany | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) (With Pembrolizumab)
Description: PFS is defined as the time from randomization until the occurrence of documented disease progression by the BICR, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria, or death from any cause in the absence of BICR-documented progressive disease.
Time Frame: Baseline to Progressive Disease or Death from Any Cause Up to 31 Months
Population: Intent to Treat (ITT) Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment. Participants censored: TRT A: 80, TRT B: 34.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Selpercatinib (TRT A): 160 mg Selpercatinib administered orally, BID continuously in 21-day cycles.
- Pemetrexed and Platinum With Pembrolizumab (TRT B): Pemetrexed 500 mg/m2, IV on Day 1 Q3W plus investigator's choice of carboplatin AUC 5 (maximum dose 750 mg) IV or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Months | 24.84 [16.89 to NA] — Upper limit of 95% confidence interval is not evaluable due to high censoring. | 11.17 [8.77 to 16.76]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With Pembrolizumab (TRT B); Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.465, 95% CI 2-sided [0.309 to 0.699]

2. Primary Outcome: PFS by BICR (With or Without Pembrolizumab)
Description: as for outcome 1
Time Frame: Baseline to Progressive Disease or Death from Any Cause Up to 31 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Participants censored: TRT A: 98, TRT B:45.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pemetrexed and Platinum With or Without Pembrolizumab (TRT B): Pemetrexed 500 mg/m2, IV on Day 1 Q3W, plus investigator's choice of carboplatin AUC 5 (maximum dose 750 mg] IV) or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 159 | 102
Months | 24.84 [17.31 to NA] — Upper limit of 95% confidence interval is not evaluable due to high censoring. | 11.17 [8.77 to 16.76]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With or Without Pembrolizumab (TRT B); Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.482, 95% CI 2-sided [0.331 to 0.700]

3. Secondary Outcome: Percentage of Participant With Disease Control Rate (DCR) by BICR (With Pembrolizumab)
Description: DCR by BICR (with Pembrolizumab) is defined as the number of participants who achieve a BOR of complete response (CR), partial response (PR), or stable disease (SD) lasting 16 or more weeks divided by the total number of participants randomized to each treatment arm.
Time Frame: Baseline to Progressive Disease or Death from Any Cause Up to 31 Months
Population: ITT Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Percentage of Participants | 89.1 [82.5 to 93.9] | 84.3 [74.7 to 91.4]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With Pembrolizumab (TRT B); Test type: Superiority; p = 0.3996, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.7 to 3.4]

4. Secondary Outcome: Percentage of Participant With DCR by BICR (With or Without Pembrolizumab)
Description: DCR by BICR (with or without Pembrolizumab) is defined as the number of participants who achieve a BOR of CR, PR, or SD lasting 16 or more weeks divided by the total number of participants randomized to each treatment arm.
Time Frame: Baseline to Progressive Disease or Death from Any Cause Up to 31 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Pemetrexed and Platinum With or Without Pembrolizumab (TRT B): Pemetrexed 500 mg/m2, IV on Day 1 Q3W plus investigator's choice of carboplatin AUC 5 (maximum dose 750 mg) IV or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 159 | 102
Percentage of Participants | 89.3 [83.4 to 93.7] | 82.4 [73.6 to 89.2]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With or Without Pembrolizumab (TRT B); Test type: Superiority; p = 0.1390, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.9 to 3.6]

5. Secondary Outcome: PFS2 (With Pembrolizumab)
Description: PFS2 is defined as the time from randomization to disease progression on the next line of treatment or death from any cause in the absence of observed disease progression.
Time Frame: Baseline to Second Disease Progression or Death from Any Cause Up to 38 Months
Population: ITT Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment. Participants censored: TRT A: 103; TRT B: 62
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pemetrexed and Platinum With Pembrolizumab (TRT B): Pemetrexed 500 mg/m2, IV on Day 1 Q3W plus investigator's choice of carboplatin AUC 5 (maximum dose 750 mg] IV) or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Months | NA [NA to NA] — Data not available due to high censoring. | NA [NA to NA] — Data not available due to high censoring.

6. Secondary Outcome: PFS2 (With or Without Pembrolizumab)
Description: as for outcome 5
Time Frame: Baseline to Second Disease Progression or Death from Any Cause Up to 38 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Participants censored: TRT A: 126; TRT B: 77
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 159 | 102
Months | NA [NA to NA] — Data not available due to high censoring. | NA [NA to NA] — Data not available due to high censoring.

7. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR) by BICR (With Pembrolizumab)
Description: ORR is defined as the number of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the total number of participants randomized to each treatment arm.
Time Frame: Baseline through Disease Progression or Death Up to 31 Months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Percentage of participants | 83.7 [76.2 to 89.6] | 65.1 [53.8 to 75.2]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With Pembrolizumab (TRT B); Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.7, 95% CI 2-sided [1.4 to 5.1]

8. Secondary Outcome: ORR: Percentage of Participants With CR or PR by BICR (With or Without Pembrolizumab)
Description: as for outcome 7
Time Frame: Baseline through Disease Progression or Death Up to 31 Months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 159 | 102
Percentage of Participants | 83.6 [77.0 to 89.0] | 62.7 [52.6 to 72.1]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With or Without Pembrolizumab (TRT B); Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.6 to 5.2]

9. Secondary Outcome: Duration of Response (DoR) by BICR (With Pembrolizumab)
Description: DoR was defined as the time from the date that measurement criteria for CR or PR (whichever is first recorded) were first met until the first date that disease was recurrent or documented disease progression was observed, or the date of death from any cause in the absence of documented disease progression or recurrence. The DOR according to both BICR and investigator-assessed BOR was evaluated per RECIST 1.1 criteria.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause Up to 31 Months
Population: ITT Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment. Participants censored: TRT A:74; TRT B: 25.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 108 | 54
Months | 24.18 [17.94 to NA] — Upper limit of 95% confidence interval not available due to high censoring. | 11.47 [9.66 to 23.26]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With Pembrolizumab (TRT B); Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.377, 95% CI 2-sided [0.224 to 0.633]

10. Secondary Outcome: DOR by BICR (With or Without Pembrolizumab)
Description: as for outcome 9
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause Up to 31 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Participants censored: TRT A: 90; TRT B: 33.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 133 | 64
Months | 24.18 [17.94 to NA] — Upper limit of 95% Confidence Interval unavailable due to high censoring. | 11.99 [9.69 to 23.26]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With or Without Pembrolizumab (TRT B); Test type: Superiority; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.418, 95% CI 2-sided [0.256 to 0.684]

11. Secondary Outcome: Overall Survival (OS) (With Pembrolizumab)
Description: Overall survival was defined as the time from randomization until death from any cause. If the participant was alive or lost to follow-up at the time of data analysis, OS data was censored on the last date the participant is known to be alive.
Time Frame: Baseline to Date of Death from Any Cause Up to 38 Months
Population: ITT Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment. Participants censored: TRT A: 104; TRT B: 68.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Months | NA [NA to NA] — Median OS data not available due to high censoring. | NA [NA to NA] — Median OS data not available due to high censoring.

12. Secondary Outcome: OS (With or Without Pembrolizumab)
Description: Overall survival was defined as the time from randomization until death from any cause. If the participant was alive or lost to follow-up at the time of data analysis, OS data will be censored on the last date the participant is known to be alive.
Time Frame: Baseline to Date of Death from Any Cause Up to 38 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Participants censored: TRT A: 127; TRT B: 84.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Selpercatinib: 160 mg Selpercatinib administered orally BID continuously in 21-day cycles.
- Pemetrexed and Platinum With or Without Pembrolizumab: Pemetrexed 500 mg/m2, IV on Day 1 Q3W plus investigator's choice of carboplatin (AUC 5 [maximum dose 750 mg] IV) or cisplatin 75mg/m2, IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib | Pemetrexed and Platinum With or Without Pembrolizumab
Number analyzed (Participants) | 159 | 102
Months | 33.05 [33.05 to NA] — Upper limit of 95% Confidence Interval unavailable due to high censoring. | NA [NA to NA] — Data not available due to high censoring.

13. Secondary Outcome: Intracranial ORR: Percentage of Participants With Intracranial CR or PR Per RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 by BICR (With Pembrolizumab)
Description: Intracranial ORR: Percentage of Participants with Intracranial CR or PR per RECIST 1.1 by BICR (with Pembrolizumab)
Time Frame: Baseline through Central Nervous System (CNS) Progression or Death up to 31 Months
Population: CNS Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment who had baseline CNS assessment and who had CNS metastasis at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 21 | 21
Percentage of participants | 81 [58.1 to 94.6] | 57.1 [34.0 to 78.2]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With Pembrolizumab (TRT B); Test type: Superiority; p = 0.1809, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.2, 95% CI 2-sided [0.8 to 12.8]

14. Secondary Outcome: Intracranial ORR: Percentage of Participants With Intracranial CR or PR Per RECIST 1.1 by BICR (With or Without Pembrolizumab)
Description: Intracranial ORR: Percentage of Participants with Intracranial CR or PR per RECIST 1.1 by BICR (with or without Pembrolizumab)
Time Frame: Baseline through CNS Progression or Death Up to 31 Months
Population: CNS Overall: All participants included in the ITT population who had baseline CNS assessment and who had CNS metastasis at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 25 | 26
Percentage of participants | 84.0 [63.9 to 95.5] | 50.0 [29.9 to 70.1]
Statistical Analysis 1: Comparison: Selpercatinib (TRT A) vs Pemetrexed and Platinum With or Without Pembrolizumab (TRT B); Test type: Superiority; p = 0.0167, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.2, 95% CI 2-sided [1.4 to 19.6]

15. Secondary Outcome: Median Intracranial DOR Per RECIST 1.1 by BICR (With Pembrolizumab)
Description: Intracranial DOR per RECIST 1.1 by BICR (with Pembrolizumab)
Time Frame: Date of Intracranial CR or PR to Date of CNS Progression or Death Due to Any Cause Up to 31 Months
Population: CNS Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment who had baseline CNS assessment and who had CNS metastasis at baseline. Participants censored: TRT A: 13; TRT B: 9.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 17 | 12
Months | NA [14.75 to NA] — Median and upper limit of 95% Confidence Interval unavailable due to high censoring. | NA [8.74 to NA] — Median and upper limit of 95% Confidence Interval unavailable due to high censoring.

16. Secondary Outcome: Median Intracranial DOR Per RECIST 1.1 by BICR (With or Without Pembrolizumab)
Description: Median Intracranial DOR per RECIST 1.1 by BICR (with or without Pembrolizumab)
Time Frame: Date of Intracranial CR or PR to Date of CNS Progression or Death Due to Any Cause Up to 31 Months
Population: CNS Overall: All participants included in the ITT population who had baseline CNS assessment and who had CNS metastasis at baseline. Participants censored: TRT A: 15; TRT B: 9.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 21 | 13
Months | NA [9.53 to NA] — Upper limit of 95% Confidence Interval unavailable due to high censoring. | 13.40 [4.17 to NA] — Upper limit of 95% Confidence Interval unavailable due to high censoring.

17. Secondary Outcome: Time to Deterioration of Pulmonary Symptoms (With Pembrolizumab)
Description: Time to Deterioration of Pulmonary Symptoms Measured by the NSCLC-Symptom Assessment Questionnaire (SAQ) (with Pembrolizumab)
Time Frame: Baseline to Deterioration of Pulmonary Symptoms Up to 31 Months
Population: ITT Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment. Participants censored: TRT A: 99; TRT B: 47.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 129 | 83
Months | NA [NA to NA] — Data not available due to high censoring. | 1.9 [0.7 to 6.6]

18. Secondary Outcome: Time to Deterioration of Pulmonary Symptoms (With or Without Pembrolizumab)
Description: Time to Deterioration of Pulmonary Symptoms Measured by the NSCLC-SAQ (with or without Pembrolizumab)
Time Frame: Baseline to Deterioration of Pulmonary Symptoms Up to 31 Months
Population: ITT Population: All randomized participants, even if a participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Participants were analyzed according to the treatment arm they were assigned to regardless of what actual treatment they received. Participants censored: TRT A: 121; TRT B: 58.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 159 | 102
Months | NA [NA to NA] — Data not available due to high censoring. | 1.6 [0.7 to 4.9]

19. Secondary Outcome: The Concordance of the Local Lab and the Central Lab RET Results: Percentage of Participants With RET-Positive Specimens as Called by the Central Lab, Which is Also RET-Positive as Called by a Local Lab (Positive Percent Agreement)
Description: The Concordance of the Local Lab and the Central Lab RET Results: Percentage of Participants with RET-Positive Specimens as Called by the Central Lab, which is also RET-Positive as Called by a Local Lab (Positive Percent Agreement)
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-06

20. Secondary Outcome: Median Time to CNS Progression Per RECIST 1.1 by BICR (With Pembrolizumab)
Description: Time to CNS Progression per RECIST 1.1 by BICR (with Pembrolizumab)
Time Frame: Baseline through CNS Progression or Death Up to 31 Months
Population: CNS Pembrolizumab: Participants included in the ITT population who were stratified with the intent to receive pembrolizumab in the event of the control-arm assignment who had baseline CNS assessment and who had CNS metastasis at baseline. Number of participants censored: TRT A = 112; TRT B = 59.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With Pembrolizumab (TRT B)
Number analyzed (Participants) | 120 | 72
Months | NA [NA to NA] — Data not available due to high censoring. | NA [NA to NA] — Data not available due to high censoring.

21. Secondary Outcome: Median Time to CNS Progression Per RECIST 1.1 by BICR (With or Without Pembrolizumab)
Description: Time to CNS Progression per RECIST 1.1 by BICR (with or without Pembrolizumab)
Time Frame: Baseline through CNS Progression or Death Up to 31 Months
Population: CNS Overall: All participants included in the ITT population who had baseline CNS assessment and who had CNS metastasis at baseline. Participants censored: TRT A: 137; TRT B: = 73.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Selpercatinib (TRT A) | Pemetrexed and Platinum With or Without Pembrolizumab (TRT B)
Number analyzed (Participants) | 146 | 88
Months | NA [NA to NA] — Data not available due to high censoring. | NA [NA to NA] — Data not available due to high censoring.

22. Secondary Outcome: Intracranial ORR: Percentage of Participants With Intracranial CR or PR Per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) by BICR (With Pembrolizumab)
Description: Intracranial ORR: Percentage of Participants with Intracranial CR or PR per RANO-BM by BICR (with Pembrolizumab)
Time Frame: Baseline through CNS Progression or Death Up to 31 Months
Reporting Status: Not Posted, anticipated posting 2026-06

23. Secondary Outcome: Intracranial ORR: Percentage of Participants With Intracranial CR or PR Per RANO-BM by BICR (With or Without Pembrolizumab)
Description: Intracranial ORR: Percentage of Participants with Intracranial CR or PR per RANO-BM by BICR (with or without Pembrolizumab)
Time Frame: Baseline through CNS Progression or Death Up to 31 Months
Reporting Status: Not Posted, anticipated posting 2026-06

24. Secondary Outcome: Intracranial DOR Per RANO-BM by BICR (With Pembrolizumab)
Description: Intracranial DOR per RANO-BM by BICR (with Pembrolizumab)
Time Frame: Date of Intracranial CR or PR to Date of CNS Progression or Death Due to Any Cause Up to 31 Months
Reporting Status: Not Posted, anticipated posting 2026-06

25. Secondary Outcome: Intracranial DOR Per RANO-BM by BICR (With or Without Pembrolizumab)
Description: Intracranial DOR per RANO-BM by BICR (with or without Pembrolizumab)
Time Frame: Date of Intracranial CR or PR to Date of CNS Progression or Death Due to Any Cause Up to 31 Months
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Baseline Up to 38 Months
Description: Safety population is defined as all participants who received study drug regardless of strata and as pre-specified, adverse events were collected for the TRT B treatment arm as a whole. Analysis of safety data will be based on the actual treatment a participant received on the first study treatment administration regardless of which treatment they were randomized to receive ("as treated").
Groups:
- Selpercatinib (TRT A): 160 milligram (mg) Selpercatinib administered orally, twice daily (BID continuously in 21-day cycles.
- Carboplatin or Cisplatin+Pemetrexed+/-Pembrolizumab (TRT B): Pemetrexed 500 milligrams per meter squared (mg/m2) administered intravenously (IV) on Day 1, every 3 weeks (Q3W), plus at the investigator's choice of carboplatin area under the concentration versus time curve 5 (AUC 5 [maximum dose 750 mg]) IV, or cisplatin 75mg/m2 IV on Day 1 Q3W for 4 cycles, plus investigator's choice with or without 200 mg pembrolizumab IV on Day 1 Q3W up to 35 cycles.
Arm/Group | Selpercatinib (TRT A) | Carboplatin or Cisplatin+Pemetrexed+/-Pembrolizumab (TRT B)
All-Cause Mortality (participants affected / at risk) | 32/158 | 17/98
Serious Adverse Events (participants affected / at risk) | 55/158 | 23/98
Other Adverse Events (participants affected / at risk) | 156/158 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selpercatinib (TRT A) (N=158) | Carboplatin or Cisplatin+Pemetrexed+/-Pembrolizumab (TRT B) (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (3)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (7) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 0 (0)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 2 (5) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (12)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selpercatinib (TRT A) (N=158) | Carboplatin or Cisplatin+Pemetrexed+/-Pembrolizumab (TRT B) (N=98)
Anaemia (Blood and lymphatic system disorders) | 18 (35) | 57 (209)
Leukopenia (Blood and lymphatic system disorders) | 11 (22) | 8 (37)
Neutropenia (Blood and lymphatic system disorders) | 6 (13) | 18 (61)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (17) | 10 (20)
Hyperthyroidism (Endocrine disorders) | 4 (8) | 7 (7)
Hypothyroidism (Endocrine disorders) | 5 (7) | 6 (10)
Lacrimation increased (Eye disorders) | 3 (5) | 13 (16)
Abdominal discomfort (Gastrointestinal disorders) | 9 (9) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 8 (11) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 18 (34) | 7 (11)
Abdominal pain upper (Gastrointestinal disorders) | 20 (31) | 13 (30)
Ascites (Gastrointestinal disorders) | 9 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 34 (46) | 39 (67)
Diarrhoea (Gastrointestinal disorders) | 69 (218) | 24 (33)
Dry mouth (Gastrointestinal disorders) | 61 (73) | 6 (6)
Nausea (Gastrointestinal disorders) | 20 (26) | 43 (93)
Stomatitis (Gastrointestinal disorders) | 19 (28) | 9 (13)
Vomiting (Gastrointestinal disorders) | 20 (38) | 23 (35)
Asthenia (General disorders) | 20 (53) | 25 (73)
Chest pain (General disorders) | 8 (9) | 13 (15)
Face oedema (General disorders) | 12 (14) | 4 (4)
Fatigue (General disorders) | 24 (40) | 26 (47)
Malaise (General disorders) | 8 (9) | 5 (8)
Oedema (General disorders) | 9 (16) | 8 (10)
Oedema peripheral (General disorders) | 41 (57) | 13 (15)
Pyrexia (General disorders) | 21 (39) | 22 (41)
Hepatic function abnormal (Hepatobiliary disorders) | 10 (41) | 1 (3)
Conjunctivitis (Infections and infestations) | 3 (3) | 5 (15)
Covid-19 (Infections and infestations) | 30 (34) | 18 (18)
Nasopharyngitis (Infections and infestations) | 9 (15) | 5 (9)
Paronychia (Infections and infestations) | 9 (10) | 0 (0)
Pneumonia (Infections and infestations) | 10 (14) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 3 (3)
Urinary tract infection (Infections and infestations) | 14 (24) | 4 (4)
Alanine aminotransferase increased (Investigations) | 95 (324) | 39 (108)
Aspartate aminotransferase increased (Investigations) | 97 (322) | 39 (94)
Bilirubin conjugated increased (Investigations) | 19 (54) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 20 (36) | 8 (12)
Blood bilirubin increased (Investigations) | 59 (230) | 1 (1)
Blood creatinine increased (Investigations) | 36 (76) | 15 (38)
Blood thyroid stimulating hormone increased (Investigations) | 10 (14) | 6 (8)
Electrocardiogram qt prolonged (Investigations) | 32 (58) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 20 (56) | 10 (15)
Lymphocyte count decreased (Investigations) | 7 (21) | 6 (28)
Neutrophil count decreased (Investigations) | 31 (126) | 25 (90)
Platelet count decreased (Investigations) | 32 (92) | 18 (46)
Weight decreased (Investigations) | 10 (31) | 9 (11)
Weight increased (Investigations) | 23 (44) | 7 (20)
White blood cell count decreased (Investigations) | 32 (142) | 25 (72)
Decreased appetite (Metabolism and nutrition disorders) | 27 (35) | 33 (56)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (8) | 9 (17)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (15) | 6 (20)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 23 (63) | 6 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (34) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (33) | 8 (25)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (24) | 5 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (47) | 6 (10)
Hypoproteinaemia (Metabolism and nutrition disorders) | 8 (24) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (22) | 12 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (16) | 6 (8)
Dizziness (Nervous system disorders) | 11 (12) | 8 (13)
Dysgeusia (Nervous system disorders) | 8 (10) | 12 (22)
Headache (Nervous system disorders) | 22 (30) | 10 (13)
Insomnia (Psychiatric disorders) | 10 (10) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 15 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 14 (18)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (12) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 8 (11) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (27) | 22 (26)
Rash (Skin and subcutaneous tissue disorders) | 35 (54) | 21 (30)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (16) | 5 (7)
Hypertension (Vascular disorders) | 76 (167) | 7 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04194944/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT04194944/SAP_001.pdf